CLINICAL TRIAL: NCT05055375
Title: The Psychology of Chinese Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Ma Fei，MD (Other)
Responsible Party: Sponsor-Investigator, Ma Fei，MD, Deputy Director of Medical Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Other Study IDs: NCC1867
Record Dates: First submitted 2018-10-22; First posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire survey — We will conduct a questionnaire survey of outpatients.

SUMMARY:
Earlier diagnosis of breast cancer in women and the use of systemic adjuvant therapy have increased the likelihood of long term, disease free survival.women who remain free of breast cancer seem to have levels of functioning and quality of life that are comparable to those of the general female population.It will be assessed the psychology status of women with breast cancer using a clinical interview,

DETAILED DESCRIPTION:
It conducts a questionnaire survey of 300 patients. The questionnaires used are: Psychological Pain Thermometer DT, Hospital Anxiety and Depression Scale HADS, Quality of Life Scale for Breast Cancer Patients FACT-B, Social Support Rating Scale SSRS. Caregivers should fill in the following scales: Psychological Pain Thermometer DT, Hospital Anxiety and Depression Scale HADS, Caregiver Burden Assessment Scale ZBI. Inclusion criteria: 1,female patients with early breast cancer after surgery; 2,no previous mental and psychological abnormalities; 3,Postoperative and prepare to accept adjuvant chemotherapy ; 4,Patient's know her/his illness .

To explore:

1. Psychological status and dynamic changes of patients and caregivers during adjuvant chemotherapy after breast cancer surgery in China.
2. The influence of psychological status of Chinese breast cancer patients on adverse reactions during adjuvant chemotherapy.
3. Gene susceptibility to psychological abnormalities during adjuvant chemotherapy for breast cancer in China.

ELIGIBILITY:
Inclusion Criteria:

Age：18~75 years; Early stage breast cancer confirmed by histology examination; Patients had undergone surgery for breast cancer; No distant metastasis; Planned to receive recommended postoperative adjuvant chemotherapy; Voluntarily provided written informed consent.

Exclusion Criteria:

Patients already receiving neoadjuvant chemotherapy before surgery; Patients had metastatic disease at diagnosis; Patients had difficulty understanding the questionnaire or communicating in Chinese; Patients had significant psychiatric or other comorbid disease prohibiting participation; Any other researcher believes that it is not appropriate to participate in this test.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese female patients with early breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-04-25 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Psychological Distress Thermometer(DT) | through study completion, an average of 2 year
  DT uses to identify sources of distress. It uses a 0 (no distress) to 10 (extreme distress).

SECONDARY OUTCOMES:
Depression Scale (HADS) | through study completion, an average of 2 year
  HADS was divided into an anxiety subscale and a depression subscale. Each item is scored from 0 (not at all) to 3 (very much) such that total scores on each sub-scale may range from 0-21.
Social Support Rating Scale (SSRS) | through study completion, an average of 2 year
  Social support was measured by SSRS. The total score ranges from 12 to 66 points, and higher score indicates higher social support for patients.
The Functional Assessment of Cancer Therapy-Breast Cancer (FACT-B) | through study completion, an average of 2 year
  The FACT-B is a 37-item instrument evaluating QoL issues. The domain scores for physical, social/family and functional well-being range from 0 to 28, the emotional domain scores from 0 to 24 points, the breast cancer- specific subscale domain scores from 0 to 40.
Zarit Caregiver Burden Interview (ZBI) | through study completion, an average of 2 year
  ZBI Is developed as 29-item self-report scale aimed to assess the subjective burden experienced by an caregiver.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersen BL, Yang HC, Farrar WB, Golden-Kreutz DM, Emery CF, Thornton LM, Young DC, Carson WE 3rd. Psychologic intervention improves survival for breast cancer patients: a randomized clinical trial. Cancer. 2008 Dec 15;113(12):3450-8. doi: 10.1002/cncr.23969. PMID 19016270
- [Background] Antoni MH, Jacobs JM, Bouchard LC, Lechner SC, Jutagir DR, Gudenkauf LM, Blomberg BB, Gluck S, Carver CS. Post-surgical depressive symptoms and long-term survival in non-metastatic breast cancer patients at 11-year follow-up. Gen Hosp Psychiatry. 2017 Jan-Feb;44:16-21. doi: 10.1016/j.genhosppsych.2016.10.002. Epub 2016 Oct 22. PMID 28041571
- [Background] Berhili S, Kadiri S, Bouziane A, Aissa A, Marnouche E, Ogandaga E, Echchikhi Y, Touil A, Loughlimi H, Lahdiri I, El Majjaoui S, El Kacemi H, Kebdani T, Benjaafar N. Associated factors with psychological distress in Moroccan breast cancer patients: A cross-sectional study. Breast. 2017 Feb;31:26-33. doi: 10.1016/j.breast.2016.10.015. Epub 2016 Oct 28. PMID 27810696
- [Background] de Souza BF, de Moraes JA, Inocenti A, dos Santos MA, Silva AE, Miasso AI. Women with breast cancer taking chemotherapy: depression symptoms and treatment adherence. Rev Lat Am Enfermagem. 2014 Oct;22(5):866-73. doi: 10.1590/0104-1169.3564.2491. PMID 25493684
- [Background] Giese-Davis J, Waller A, Carlson LE, Groff S, Zhong L, Neri E, Bachor SM, Adamyk-Simpson J, Rancourt KM, Dunlop B, Bultz BD. Screening for distress, the 6th vital sign: common problems in cancer outpatients over one year in usual care: associations with marital status, sex, and age. BMC Cancer. 2012 Oct 2;12:441. doi: 10.1186/1471-2407-12-441. PMID 23031647
- [Background] Gold M, Dunn LB, Phoenix B, Paul SM, Hamolsky D, Levine JD, Miaskowski C. Co-occurrence of anxiety and depressive symptoms following breast cancer surgery and its impact on quality of life. Eur J Oncol Nurs. 2016 Feb;20:97-105. doi: 10.1016/j.ejon.2015.06.003. Epub 2015 Jul 15. PMID 26187660
- [Background] Gregorowitsch ML, van den Bongard HJGD, Young-Afat DA, Pignol JP, van Gils CH, May AM, Verkooijen HM. Severe depression more common in patients with ductal carcinoma in situ than early-stage invasive breast cancer patients. Breast Cancer Res Treat. 2018 Jan;167(1):205-213. doi: 10.1007/s10549-017-4495-y. Epub 2017 Sep 11. PMID 28894982
- [Background] Guo X, Xu J, Ying E, Yu Z, Sun T. Correlation between hormone receptor status and depressive symptoms in patients with metastatic breast cancer. Oncotarget. 2017 Feb 2;8(31):50774-50781. doi: 10.18632/oncotarget.15037. eCollection 2017 Aug 1. PMID 28881602
- [Background] Kaminska M, Kubiatowski T, Ciszewski T, Czarnocki KJ, Makara-Studzinska M, Bojar I, Staroslawska E. Evaluation of symptoms of anxiety and depression in women with breast cancer after breast amputation or conservation treated with adjuvant chemotherapy. Ann Agric Environ Med. 2015;22(1):185-9. doi: 10.5604/12321966.1141392. PMID 25780852
- [Background] Kim SY, Kim SW, Shin IS, Park MH, Yoon JH, Yoon JS, Kim JM. Changes in depression status during the year after breast cancer surgery and impact on quality of life and functioning. Gen Hosp Psychiatry. 2018 Jan-Feb;50:33-37. doi: 10.1016/j.genhosppsych.2017.09.009. Epub 2017 Sep 29. PMID 28987920
- [Background] Kim YH, Choi KS, Han K, Kim HW. A psychological intervention programme for patients with breast cancer under chemotherapy and at a high risk of depression: A randomised clinical trial. J Clin Nurs. 2018 Feb;27(3-4):572-581. doi: 10.1111/jocn.13910. Epub 2017 Jul 6. PMID 28557043
- [Background] Ng CG, Mohamed S, Kaur K, Sulaiman AH, Zainal NZ, Taib NA; MyBCC Study group. Perceived distress and its association with depression and anxiety in breast cancer patients. PLoS One. 2017 Mar 15;12(3):e0172975. doi: 10.1371/journal.pone.0172975. eCollection 2017. PMID 28296921
- [Background] So WK, Marsh G, Ling WM, Leung FY, Lo JC, Yeung M, Li GK. Anxiety, depression and quality of life among Chinese breast cancer patients during adjuvant therapy. Eur J Oncol Nurs. 2010 Feb;14(1):17-22. doi: 10.1016/j.ejon.2009.07.005. Epub 2009 Sep 5. PMID 19734087
- [Background] Zhang J, Zhou Y, Feng Z, Xu Y, Zeng G. Longitudinal Trends in Anxiety, Depression, and Quality of Life During Different Intermittent Periods of Adjuvant Breast Cancer Chemotherapy. Cancer Nurs. 2018 Jan/Feb;41(1):62-68. doi: 10.1097/NCC.0000000000000451. PMID 27922916